CLINICAL TRIAL: NCT03679208
Title: Safety and Performance of the Intra-articular Injection of Animal-free Chitosan Biomaterial (Viscosupplementation) in Patients With Symptomatic Knee Osteoarthritis: a Pre-market Study.
Brief Title: sAfety PerfoRmance chitOsan osteOarthritis ViscosupplEmentation
Acronym: APROOVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kiomed Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KIO014-APROOVE
Record Dates: First submitted 2018-07-09; First posted 2018-09-20 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage 1 Safety cohort (Experimental): Two injections of the investigational device (KIO014) at 3-month interval in 10 patients and 12-month follow-up to establish long-term safety as primary endpoint.
  Interventions: Device: Investigational device coded KIO014
- Stage 2 Performance (test group) (Experimental): One injection of the investigational device (KIO014) in 60 patients to evaluate the reduction in pain at 3 months as primary endpoint. Additional follow-up at 6 months.
  Interventions: Device: Investigational device coded KIO014
- Stage 2 Performance (control group) (Active Comparator): One injection of the control device (Durolane(r)) in 30 patients to evaluate the reduction in pain at 3 months as control endpoint. Additional follow-up at 6 months.
  Interventions: Device: Durolane(r) as control device

INTERVENTIONS:
Device: Investigational device coded KIO014 — Innovative chitosan-based biomaterial intended for intraarticular injection.
  Arms: Stage 1 Safety cohort; Stage 2 Performance (test group)
Device: Durolane(r) as control device — Crosslinked hyaluronic acid-based biomaterial intended for intraarticular injection.
  Arms: Stage 2 Performance (control group)

SUMMARY:
KIO014 is an innovative chitosan-based biomaterial intended for synovial fluid viscosupplementation indicated for the symptomatic treatment of knee osteoarthritis (OA). The study KIO014-APROOVE is aimed to evaluate the safety and performance of KIO014 in patients with symptomatic knee OA. A total of 100 patients will be enrolled. The study is divided in two stages. The Stage 1 cohort is the safety cohort where 10 patients will be enrolled. Stage 1 patients receiving two injections of KIO014 at day 0 and at month 3, and will be followed for 12 months post initial injection. The Stage 2 cohort is the performance cohort for 90 patients, and this stage will be randomized controlled and single-blind for the patient. In stage 2, 60 patients will receive an intra-articular injection of KIO014 (test group) and 30 patients will receive an intra-articular injection of Durolane® (control group). Patients will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with age ≥ 40 years and ≤ 85 years except in Stage 1 cohort where age is limited to ≤ 70 years.
* Body mass index (BMI) ≤ 35 kg/m².
* Uni- or bilateral femorotibial knee OA associated or not with femoropatellar knee OA.
* Primary knee osteoarthritis responding to the clinical and radiological criteria of the American College of Rheumatology (ACR)
* Radiological Kellgren and Lawrence (K&L) grade II to III from a standing knee radiograph taken less than 6 months previously.
* Symptomatic pain at least 6 months in the treatment knee not or poorly responding to first line non-opioid analgesics and non-steroidal anti-inflammatory drug in oral uptake.
* Pain criteria assessed prior to injection at visit 1 after mandatory 48-hour wash-out:

  * Treatment knee: 7-17 points of the 5-graded Likert WOMAC pain score and at least 2 points on the WOMAC pain subscore A1 in the most affected knee.
  * Non-treatment knee: not more than 6 points of the 5-graded Likert WOMAC pain score in the contralateral knee.
* Fully ambulatory patient for functional evaluation
* Willing NOT to take any pain medication for 48 hours prior to study visit.
* For female NOT surgically sterile (tubal ligation or hysterectomy) or NOT postmenopausal for at least one year, must have an effective contraception (pill, patch, ring, diaphragm, implant and intrauterine device).
* Able to understand and follow the instructions of the study.
* Having signed a written informed consent.

Exclusion Criteria:

* Related to the OA pathology and related symptoms:

  * Radiological K&L grade 0, I or IV from a standing knee radiograph taken less than 6 months previously.
  * Exclusively patellofemoral osteoarthritis where the symptoms, including pain, are principally of patellofemoral origin (Patellar syndrome).
  * Chondromatosis or villonodular synovitis of the knee.
  * Clinically-apparent knee effusion, inflammation or flare-up of the knee or abnormal synovial fluid macroscopy or volume upon arthrocentesis on the day of injection.
  * History of injury to the treatment knee during the 6 months before inclusion or recent trauma (<1 month) of the knee responsible of pain that is not directly related to OA symptoms.
  * Significant clinically-assessed or radiographic varus or valgus deformation of the selected knee at the judgment of the investigator.
  * Inflammatory disease.
  * Pathologies interfering with the evaluation of OA pain for the knee to be treated.
* Related to treatments:

  * Contraindications: hypersensitivity or allergy to the product components of KIO014, including chitosan, sorbitol and/or other mushroom-derived products, or to hyaluronic acid-based products.
  * Corticosteroids or Plasma Rich Platelet (PRP) or cell-based therapy injection in the treatment knee in the last 3 months before injection.
  * Hyaluronic acid injection in the treatment knee in the last 6 months before injection.
  * Arthroscopy and surgery in the treatment knee in the last 6 months before injection.
  * Oral corticotherapy ≥5 mg/day (in prednisone equivalent) in the last 3 months before injection.
  * Change in the dosage regimen of symptomatic slow-acting drugs (SYSAD) or dietary supplement in the last 3 months before injection.
  * Change in physiotherapy of the treatment knee in the last 3 months.
  * Anticipated need for any surgical or other invasive procedure during the trial including prosthesis in the treatment knee.
  * Anticipated need for any forbidden OA treatments during the trial except for rescue treatment as defined in the study protocol.
  * Anticoagulants: coumarin-based compounds or heparin.
* Related to associated diseases:

  * Any Investigator-assessed clinically significant condition that may represent a substantial risk to the patient or may have an impact on the study assessments.
  * History of recurrent bacterial infection, defined as at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years or history of synovial infection or infections or skin diseases in the area of the injection site.
  * History of symptomatic hip OA
  * History of autoimmune disease.
  * Severe, ongoing and uncontrolled diseases, or other major disease, or other severe uncontrolled conditions.
  * Subject addicted to alcohol or drugs or ongoing or recently recovered depression or psychiatric disorders or any other disorder and/or that may pose a health risk to the subject in the study and/or may have an impact on the study assessments.
  * Severe alteration of mobility preventing any functional evaluation.
  * High risk of hemorrhage.
* Related to patients:

  * Participation in a therapeutic clinical trial in the last 3 months before injection.
  * Patient under guardianship or judicial protection.
  * Pregnancy, breastfeeding, planned conception, or premenopausal women without effective contraception, tubal ligation or hysterectomy.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-05-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety using 4-point numerical rating scale for local effects | All time points for up to 12 months
  At each visit, the treatment knee is assessed for the occurrence of local effects (joint pain, effusion or swelling) using a 4-point numerical rating scale (NRS) graded 0-3 (none, mild, moderate or severe).
Change in pain at 3 months versus pre-injection baseline using the 5-graded Likert self-administered WOMAC pain questionnaire (Stage 2 cohort only) | 3 months
  The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a self-administered questionnaire designed to assess pain, stiffness, and physical function through a series of 24 questions divided into 3 subscales. The WOMAC pain score consists of 5 questions. Each question is graded 0-4 on the 5-graded Likert scale (none, mild, moderate, severe or extreme) relating to how much pain the subject has experienced during the last 48 hours. The mean score is reported.

SECONDARY OUTCOMES:
Changes from baseline in total score, pain, stiffness, and physical functioning subscales of the treatment knee as measured using the 5-graded Likert WOMAC at the different time points over 6 months. | 6 months
  The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a self-administered questionnaire designed to assess pain, stiffness, and physical function through a series of 24 questions divided into 3 subscales. Each question is graded 0-4 on the 5-graded Likert scale (none, mild, moderate, severe or extreme) relating to how much pain, stiffness or daily physical activities the subject has experienced during the last 48 hours. The score of each dimension, namely pain, stiffness and physical function, is calculated by simply adding the score for each question using the 5-graded Likert scale from 0 to 4. For each dimension, the mean score is reported.
Changes from baseline in subject's pain using an 11-point Numerical Rating Scale (NRS) at the different time points over 6 months. | 6 months
  Pain at rest is evaluated using a self-administered 11-point numerical rating scale (NRS) from "no pain = 0" to "worst pain = 10". Subject's pain can be used as a criterion for evaluating the OMERACT-OARSI responders.
Changes from baseline in subject's global assessment using an 11-point Numerical Rating Scale (NRS) at the different time points over 6 months. | 6 months
  Subject's global assessment is evaluated using a self-administered 11-point numerical rating scale (NRS) from "very poor = 0" to "excellent = 10". Subject's global assessment can be used as a criterion for evaluating the OMERACT-OARSI responders.
Response to treatment according to Osteoarthritis Research Society International (OARSI) Standing Committee for Clinical Trials Response Criteria Initiative and the Outcome Measures in Rheumatology (OMERACT) at the different time points over 6 months. | 6 months
  The proportion of subjects meeting the OMERACT criteria for the response to treatment from the Osteoarthritis Research Society International (OARSI) Standing Committee for Clinical Trials Response Criteria Initiative and the Outcome Measures in Rheumatology (OMERACT).
Treatment responders with >40% improvement in pre-injection pain (WOMAC Likert) at the different time points over 6 months. | 6 months
  The proportion of subjects with a 40% improvement in pre-injection pain as evaluated by the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) pain score using the 5-graded Likert scale from 0 to 4 (none, mild, moderate, severe or extreme) relating to how much pain the patient has experienced during the last 48 hours.